CLINICAL TRIAL: NCT06811051
Title: Effects of Clove Oil and Menthol-containing Lozenges in Preventing Post-extubation Sore Throat in Patients Undergoing Surgical Intervention
Brief Title: Effect of Clove Oil and Menthol Lozenges on Post-extubation Sore Throat
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Atlas University (Other)
Collaborators: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Cagla Toprak, Atlas University, Atlas University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CToprak
Record Dates: First submitted 2025-01-08; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-02

CONDITIONS: Sore Throat
Keywords: sore throat; lozenge; postoperative
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Menthol Group Patients (Experimental): Patients in the menthol group will fill out the Patient introduction form, patient follow-up form, and numerical pain scale just before the first application. After 60 minutes after extubation, they will be asked to take the lozenge into their mouth without chewing or swallowing it and suck it, and the patient will be monitored until the lozenge is completely dissolved. After the first lozenge is finished, the patient follow-up form and numerical pain scale will be filled out. The second lozenge will be sucked 90 minutes after extubation. The third lozenge will be sucked 120 minutes after extubation and the patient follow-up form and numerical pain scale will be filled out.
  Interventions: Biological: Menthol lozenge
- Clove lozenge group (Experimental): Patients in the clove group will fill out the Patient introduction form, patient follow-up form, and numerical pain scale just before the first application. After 60 minutes after extubation, they will be asked to take the lozenge into their mouth without chewing or swallowing it and suck it, and the patient will be monitored until the lozenge is completely dissolved. After the first lozenge is finished, the patient follow-up form and numerical pain scale will be filled out. The second lozenge will be sucked 90 minutes after extubation. The third lozenge will be sucked 120 minutes after extubation and the patient follow-up form and numerical pain scale will be filled out.
  Interventions: Biological: Clove lozenge
- Control Group (Placebo Comparator): Before routine clinical procedures after surgery, the patients in the control group will fill out the Patient introduction form, Patient follow-up form, and Numerical pain scale. After 60 minutes after extubation; clinical procedures do not include any procedures or interventions and the patient follow-up form and Numerical pain scale will be evaluated. After 120 minutes after extubation; the patient follow-up form and numerical pain scale will be evaluated.
  Interventions: Other: None-placebo

INTERVENTIONS:
Biological: Menthol lozenge — Patients in the menthol group will fill out the Patient introduction form, patient follow-up form, and numerical pain scale just before the first application. After 60 minutes after extubation, they will be asked to take the lozenge into their mouth without chewing or swallowing it and suck it, and the patient will be monitored until the lozenge is completely dissolved. After the first lozenge is finished, the patient follow-up form and numerical pain scale will be filled out. The second lozenge will be sucked 90 minutes after extubation. The third lozenge will be sucked 120 minutes after extubation and the patient follow-up form and numerical pain scale will be filled out.
  Arms: Menthol Group Patients
Biological: Clove lozenge — Patients in the clove group will fill out the Patient introduction form, patient follow-up form, and numerical pain scale just before the first application. After 60 minutes after extubation, they will be asked to take the lozenge into their mouth without chewing or swallowing it and suck it, and the patient will be monitored until the lozenge is completely dissolved. After the first lozenge is finished, the patient follow-up form and numerical pain scale will be filled out. The second lozenge will be sucked 90 minutes after extubation. The third lozenge will be sucked 120 minutes after extubation and the patient follow-up form and numerical pain scale will be filled out.
  Arms: Clove lozenge group
Other: None-placebo — Before routine clinical procedures after surgery, the patients in the control group will fill out the Patient introduction form, Patient follow-up form, and Numerical pain scale. After 60 minutes after extubation; clinical procedures do not include any procedures or interventions and the patient follow-up form and Numerical pain scale will be evaluated. After 120 minutes after extubation; the patient follow-up form and numerical pain scale will be evaluated.
  Arms: Control Group

SUMMARY:
In patients undergoing surgical intervention, endotracheal intubation, which is a part of the anesthesia procedure, can cause postoperative sore throat in patients. This situation causes difficulty in swallowing, inadequate nutrition and fluid intake, and prolongs the recovery process. In addition, sore throat is defined as a source of physical stress, which can lead to an increase in the incidence of postoperative morbidity and a decrease in patient satisfaction. This study aimed to investigate the effect of menthol and clove oil lozenges on sore throat after surgery. Our aim was to provide evidence on the effectiveness of simple, low-cost menthol and clove oil lozenges in reducing sore throat after extubation, thus helping the patient recover.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of menthol and clove oil lozenges on sore throat in patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65. Having had abdominal surgery. Being extubated within the first 8 hours after surgery. ASA class I-III. Mallampati class I-II. Glasgow Coma Scale (GCS) score 15

Exclusion Criteria:

* History of allergies.

  * Severe nausea and vomiting.
  * Being extubated after the first 8 hours after surgery.
  * Communication disorders
  * Mallampati class III-IV.
  * Glasgow Coma Scale (GCS) score <15

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
VAS pain score | Pain was assessed at 4 time points, immediately before the first application (baseline) and 30 minutes after application of each of the three lozenges (T1, T2, T3).
  Sore throat pain will be measured by VAS score: zero mean NO PAIN, 10 means unsupportable pain.
sore throat | 60 minutes after extubation
  VAS is used to make measurable some values that cannot be measured numerically, evaluated by individuals by marking them on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end of which indicates that the individual is "very bad".

SECONDARY OUTCOMES:
Sore throat | 90 minutes after extubation
  VAS is used to make measurable some values that cannot be measured numerically, evaluated by individuals by marking them on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end of which indicates that the individual is "very bad".

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Atlas University, Istanbul, Kağıthane
  - Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: sore throat after extubation — https://pubmed.ncbi.nlm.nih.gov/?term=sore+throat+after+extubation&filter=datesearch.y_5